CLINICAL TRIAL: NCT01989975
Title: A Multi-center, Non-randomized Study in Subjects With Diabetes Mellitus Treated With Sensor-Augmented Pump Therapy to Evaluate the Performance and Safety of CareLink Connect Transferring Pump Data to Web Connected Devices Via CareLink
Brief Title: CareLink Connect - Technical Evaluation Study
Status: Completed | Type: Observational
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Other Study IDs: EUR06
Record Dates: First submitted 2013-04-22; First posted 2013-11-21 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus
Keywords: Sensor-Augmented Pump Therapy; Connected Care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the performance, patient satisfaction and safety of connectivity gateway device CareLink Connect, transferring CGM (Continuous Glucose Monitoring) data from a VEO insulin pump to CareLink online (every 5th minute) and thereby making it available for patients or Care Partners individual web connected devices such as smartphones, tablets and PCs.

ELIGIBILITY:
Inclusion Criteria:

1. Subject between the age of 12 - 65 years that has a clinical diagnosis of insulin requiring diabetes for at least 1 year
2. Subject is currently using a Paradigm® Veo™ Medtronic insulin pump for at least 3 months and willing to continue to use for the duration of the study.
3. Subject has sufficient Continuous Glucose Monitoring use experience, as determined by the Investigator, and is willing to continuously use CGM for the duration of the study.

   Guidelines to evaluate the patients experience are:

   i. Subject has a minimum of 30 days of CGM use within a year prior to enrollment.

   ii. Subject has experience with and is able to, or has a Care Partner who can:
   1. Insert/change sensor,
   2. Recharge the transmitter.
   3. Read sensor data in real-time on the insulin pump screen.
4. Subject is willing to, or has a Care Partner who can, perform at least the minimum required (2 per day) Blood Glucose readings to maintain CGM Sensor calibration.
5. Subject, if under the age of 18, has a Care Partner who is willing to participate to the study, attend the study visit with the subject, and complete user's feedback questionnaires and Care Partner diary. Care Partners are optional for patients of 18 years of age or older.
6. Subject and/or Care Partner have access to a computer with Internet access.
7. Subject and/or Care Partner have access to an Internet connected device.
8. Subject, or their legal guardian, is willing to allow a Care Partner to receive and view information transmitted by their Paradigm® Veo™ Medtronic insulin pump to a Mobile phone/Smartphone/tablet/PC via the CareLink Connect/CareLink Personal System.
9. Subject is willing to keep CareLink Connect device in the same room as themselves or regularly carry the study device with them and maintain its operational status (at approximately 16h per 24h).
10. Subject is willing to keep a short diary during the device use reporting time periods away(for more than one hour) from the CareLink Connect device.
11. Subject is in good general health as judged by the PI.

Exclusion Criteria:

1. Female subject is pregnant, per urine pregnancy test performed at screening in women of child-bearing potential
2. Female subject plans to become pregnant during the course of the study
3. Subject is unable to tolerate tape adhesives of the infusion set and CGM sensor
4. Subject has any unresolved adverse skin condition in the area of the pump infusion set or the CGM sensor placement (e.g. psoriasis, rash, Staphylococcus infection)
5. The subject has known cellular connectivity problem at their home
6. The subject is by the PI judged ineligible or unable to perform the study procedures jeopardizing the study results.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Steno Diabetes Center, Gentofte Municipality, Denmark
- Diabeter, Rotterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetes Subjects With Sensor-Augmented Pump Therapy: Subjects with diabetes mellitus treated with Sensor-Augmented Pump therapy participated the study for 15 days
Period: Overall Study
Arm/Group | Diabetes Subjects With Sensor-Augmented Pump Therapy
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diabetes Subjects With Sensor-Augmented Pump Therapy
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 22
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 25
  Denmark | 15

OUTCOME MEASURES:

1. Primary Outcome: CareLink Connect Activity: % of the Time Per Day When Cellular Connection Was Established
Description: The overall system connectivity between the pump, the CareLink Connect device, and the CareLink server will be measured. CareLink Connect activity will be measured by:
  * Date and time of CareLink Connect transmissions
  * Transmission type and data sent in CareLink Connect transmissions (includes RF messages and history uploads)
Time Frame: Outcome measured after 15 days of use of the CareLink Connect Device
Measure: Mean (Standard Deviation); unit: percentage of time spent connected
Arm/Group | Diabetes Subjects With Sensor-Augmented Pump Therapy
Number analyzed (Participants) | 40
percentage of time spent connected | 89.3 (12.4)

2. Primary Outcome: Subject Experience After Using the Carelink Connect Device
Description: Subject experience after using the Carelink Connect device was evaluated with questionnaires. Subjects were asked the question: I felt that I had good control over my diabetes. Likert Scale of 1-7 was used in the study to evaluate the question (1 being the the worse, 4 being neutral and 7 being the best).
Time Frame: Outcome measured after 15 days of use of the CareLink Connect Device
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Diabetes Subjects With Sensor-Augmented Pump Therapy
Number analyzed (Participants) | 40
Scores on a Scale | 5.6 (1.1)

3. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Descriptive summary of number and type of serious adverse events (SAE)
Time Frame: Outcome measured after 15 days of use of the CareLink Connect Device
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Subjects With Sensor-Augmented Pump Therapy
Number analyzed (Participants) | 40
Participants | 0

4. Secondary Outcome: Number of Participants With Investigational Device Deficiencies
Description: Subjects were instructed to report any inadequacies of a medical device including:
  * Lack of connection between the CareLink Connect device and the Veo pump (Connectivity issues)
  * Device Battery issue
  * Device information display issue
Time Frame: Outcome measured after 15 days of use of the CareLink Connect Device
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Subjects With Sensor-Augmented Pump Therapy
Number analyzed (Participants) | 40
Participants
  Connectivity issues | 22
  Device battery issues | 2
  Information display issues | 4
  No Issues | 12

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Diabetes Subjects With Sensor-Augmented Pump Therapy
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 9/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetes Subjects With Sensor-Augmented Pump Therapy (N=40)
Headache (Nervous system disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Severe common cold (Infections and infestations) | 1 (1)
Minor nausea (Gastrointestinal disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Cold (Infections and infestations) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Infection external ear (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days